CLINICAL TRIAL: NCT06784921
Title: Real-World Patient Characteristics, Treatment Patterns, and Outcomes for Patients With HER2 Negative Metastatic Breast Cancer Treated With Sacituzumab Govitecan: A Retrospective Trial in China（SACIT-OUT）
Brief Title: To Investigate the Real-world Efficacy and Safety of Sacituzumab Govitecan for HER2 Negative Metastatic Breast Cancer Patients in China.
Acronym: SACIT-OUT
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Xiaojia, MD, Zhejiang Cancer Hospital
Other Study IDs: IRB-2023-1203
Record Dates: First submitted 2025-01-16; First posted 2025-01-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Metastatic
Keywords: Breast cancer; Sacituzumab Govitecan
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect puncture tissue specimens before and after drug use for proteomics detection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the real-world efficacy and safety of Sacituzumab govitecan for HER2 negative metastatic breast cancer patients in China.

DETAILED DESCRIPTION:
This study will conduct a multicenter, open, prospective clinical trial to investigate the real-world efficacy and safety of Sacituzumab govitecan for HER2 negative metastatic breast cancer patients in China.

ELIGIBILITY:
Inclusion Criteria:

Local recurrent or metastatic breast cancer suitable for chemotherapy, confirmed histologically.

HER2-negative breast cancer(according to 2018 ASCO/CAP HER2 test guideline). 18-75 years old. ECOG PS 0～2. life expectancy is not less than 12 weeks. at least one measurable lesion according to RECIST 1.1. received at least two cycles of SG. Signed informed

Exclusion Criteria:

Patients who did not receive sacituzumab govitecan treatment for two or more cycles Other malignant tumors, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma, have been diagnosed in the past five years.

Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial History of neurological or psychiatric disorders Researchers believe that patients are not suitable for any other situation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient had a diagnosis of metastatic breast cancer, received at least two cycles of sacituzumab govitecan.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | from enrollment to progression or death (for any reason),assessed up to 100 months
  Progression-Free Survival

SECONDARY OUTCOMES:
Objective Response Rate | from enrollment to progression or death (for any reason), assessed up to 100 months
  Ratio of CR and PR in all subjects
DoR | The first evaluation of CR or PR to progression or death (for any reason),assessed up to 100 months
  Duration of Response
OS | from enrollment to death (for any reason).assessed up to 100 months
  Overall Survival

OTHER OUTCOMES:
adverse event | from enrollment to 30 days after the last dose administrate
  Adverse events are described in terms of CTC AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojia Wang, MD; Ph.D, Principal Investigator — Zhejiang Cancer Hospital; Qin Wu, Ph.D, Principal Investigator — Hangzhou Institute of Medicine (HIM); Huanhuan Zhou, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided